CLINICAL TRIAL: NCT04648124
Title: VIsual Cerebral ConnecTivity On Functional Magnetic Resonance Imaging in Patients With Hereditary REtinal Dystrophies
Acronym: VICTOIRE
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2020_30
Record Dates: First submitted 2020-08-26; First posted 2020-12-01 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Vision Functional Brain Networks in Patients With Hereditary Retinal Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients for whom there is no planned implant surgery
  Interventions: Device: IRMf-r (séquence resting state)
- Patients for whom implantation surgery is planned
  Interventions: Device: IRMf-r (séquence resting state)
- case
  Interventions: Device: IRMf-r (séquence resting state)

INTERVENTIONS:
Device: IRMf-r (séquence resting state) — Functional MRI of functional brain networks

SUMMARY:
The Rothschild Foundation A Hospital follows a cohort of approximately 300 patients with hereditary retinal dystrophy. These patients are followed in ophthalmology consultation every year. In order to plan the MRI on the day of the annual consultation and to avoid additional travel for patients, patients will be informed of the study before the consultation (transmission of an information letter and the information note from study). If patients agree to participate in the study, rMRI will be scheduled. During the follow-up ophthalmologic consultation, after checking the inclusion and non-inclusion criteria, the study information will be repeated, and patients who still agree to participate will sign the study consent.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Diagnostic clinique de dystrophie rétinienne héréditaire ou maculopathie héréditaire, syndromique ou non syndromique
* Artificial vision treatment such as a retinal implant, or optogenetics scheduled in the next 6 months
* Express consent to participate in the study
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman
* Contraindication to MRI (claustrophobia, implanted equipment such as pacemaker).
* Other additional ocular pathology that can significantly affect vision
* Recent eye surgery less than 3 months old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hereditary retinal dystrophies whether or not to undergo implantation surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Localization and characterization of neural networks | baseline
  neuronal networks description using rest and morphological functionnal MRIs
Evolution of neuronal networks after retinal implantation | baseline
  neuronal networks description using rest and morphological functionnal MRIs

CONTACTS AND LOCATIONS:
Overall Officials: Augustin LECLER, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation Adolphe de Rothschild, Paris, PARIS, France

IPD SHARING:
Plan to Share IPD: No